CLINICAL TRIAL: NCT06646822
Title: Prevalence, Patterns, Awareness and Attitudes of Stimulant Drug Use Among Students in Egyptian Universities: a Cross-sectional Study.
Brief Title: Prevalence, Awareness, Attitudes and Patterns of Stimulant Drug Use Among Students in Egyptian Universities
Acronym: SDU
Status: Active, not recruiting | Type: Observational
Sponsor: Asmaa Ahmed Hamed Mohie Eldin (Other)
Responsible Party: Sponsor-Investigator, Asmaa Ahmed Hamed Mohie Eldin, Associate professor, New Valley University
Organization: New Valley University (Other)
Other Study IDs: MPEC 240704; MPEC 240704 (Registry Identifier: Minia University)
Record Dates: First submitted 2024-10-09; First posted 2024-10-17 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-10

CONDITIONS: Study of Stimulants in Egypt
Keywords: Prevalence; awareness; attitudes; Stimulant drug; Egyptian universities
MeSH Terms: conditions — Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group: Undergraduate students at a large public university in Egypt who were 18 years of age or older took the survey in 2024. All survey and recruitment materials were approved by Minia University, faculty of pharmacy.
  Students were received survey through email. Students took the survey online at a time and location of their choice.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — observational study

SUMMARY:
Stimulants are dangerous drugs that are commonly abused by individuals looking to stay alert and focused, lose weight, stay awake, and get high. Although these drugs can be extremely harmful and even life-threatening, many of them can also be used to treat conditions like ADHD, narcolepsy, and in some cases, depression. There are many types of stimulant drugs, and it can be beneficial to know a little about each one, its purposes, and how harmful it can be when abused.

Illicit stimulants are usually schedule II, depending on whether or not they can be used to treat medical conditions. While some variations of stimulants are schedule I drugs, most are extremely addictive and dangerous schedule II substances. These drugs are often abused in a binge-crash pattern. According to the NIDA Teen, "In order to keep the 'high' going, people may take the drug repeatedly within a short period of time, at increasingly higher doses." This makes these drugs extremely addictive.

The aim of this survey to detect prevalence of non prescription stimulants in Egyptian students and increase their awareness of the harmful effects of these drugs.

DETAILED DESCRIPTION:
Methodology Undergraduate students at a large public university in Egypt (Minia, Assuit, Souhag, South Valley) who were 18 years of age or older took the survey in 2024. All survey and recruitment materials were approved by Minia University, faculty of pharmacy.

Students will receive survey through email. Students took the survey online at a time and location of their choice. No time limit was imposed. Participants will automatically routed through each section of the survey. First, students read a description of the study, including potential benefits and costs of taking the survey, and then they will be asked if they are a current undergraduate student at the participating university and their age. First section included the demographic data of participants, the second section the investigator will aske participants to indicate if they had ever been prescribed a stimulant. If participant answered yes, participants will route to the next section which asks about the frequency of use, the effects of stimulants and any complain if present.

ELIGIBILITY:
Inclusion Criteria:

- Academic student Age (18-30) years Included in medical faculty

Exclusion Criteria:

* Not undergraduates student Aged < 18 years

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 18-30
Study Population: Undergraduate students at a large public university in Egypt who were 18 years of age or older took the survey in 2024. All survey and recruitment materials were approved by Minia University, faculty of pharmacy.
  Students were received survey through email. Students took the survey online at a time and location of their choice. No time limit was imposed.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence/ pattern | 1 year
  * - Do/ did you use stimulants ( Recreational drugs): Yes No
  * How do / did you obtain this medication Prescribed Non prescribed
  * When did you start receiving stimulants for last 1 year for last 3 years for last 5 years
  * Which Stimulant (drug) is/ was used
    * tobacco products (e.g., coffee, chocolate, cigarettes) high caffeine products
    * pseudoephedrine, ( nasal decongestant)
    * methylphenidate [Ritalin]
    * amphetamine [Adderall]
    * methamphetamine
    * modafinil (Provigil)
    * dextroamphetamine (Dexedrine)
    * dextro/levoamphetamine (Adderall)
    * adrafinil (Olmifon)
    * piracetam
    * Others
Awareness/ attitude | 1 year
  - How do you know about the effect of stimulants: Substance use by peers Friends as a source of prescription stimulants Social media Promotion
  * Why do you use stimulant Because it helps me concentrate Because it helps me study and enhance memory Because it helps increase my alertness and concentration Because it gives me a high mood Because it helps me to be more energetic Because it improves sleep quality Because it decreases stress level Because of experimentation Because it helps me lose weight
  * Do you know that stimulant is harmful to the body systems Yes No
  * Which of the following side effects do you experience after using stimulant
    * decreased appetite
    * weight loss
    * headache
    * insomnia
    * dizziness
    * nervousness.
    * Seizures
    * cardiac events (increase blood pressure and heart rate, heart attacks)
    * psychosis
  * Did you receive treatment for the side effects after using stimulants Yes No

SECONDARY OUTCOMES:
Demographic data | 1 year
  - Age: 18-20 20-22 22-25
  - Sex: Male Female
  - Residence: Rural Urban
  * University Minia Assiut South Valley Suhag
  * Faculty Pharmacy Medicine
  * Academic Year:
  First tear second year Third year fourth year Fifth year
  * Cigarette smoking Yes No
  * Associated disorder:
  psychic (e.g. ADHD)
  * income or economic level Low income moderate income high income
  * visits to emergency department or hospital (times/ year) 1-3 4-10 11-15 >15

CONTACTS AND LOCATIONS:
Locations (1):
- Asmaa Ahmed Hamed, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No